CLINICAL TRIAL: NCT06458205
Title: Population Medicine Multimorbidity Interventions in Xishui on High-risk COPD Smokers: a Cluster Randomized Controlled Trial
Brief Title: Impact of Multi-Component Interventions on High-Risk COPD Smokers
Acronym: POPMIX-Smoking
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Simiao Chen, Professor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAMS&PUMC-IEC-2024-042
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-06

CONDITIONS: Multimorbidity; Tobacco Use Cessation; Smoking Reduction
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): For all townships within the intervention arm, we have constructed a pay-for-population mechanism to incentivize all medical practitioners to care for population health within each township. For smokers, we will provide a multi-component intervention: (1) NicQuit, a CBT-based digital health intervention for those who use intelligent mobile phones; (2) community-based pulmonary function test; (3) health education and encouragement to seek medication in superior hospitals for those spirometry-defined COPD patients; (4) CBT-based health education to the abnormal BMI; (5) health education to smoking cessation; (6) Active recruitment of smokers with high blood pressure or high blood glucose measurement. Intensive follow-ups will be at month 3, 6, and 12.
  Interventions: Combination Product: Multi-component intervention for smokers
- Control Arm (No Intervention): We will notify smokers with high-risk COPD to seek further diagnoses in superior hospitals. We provide a face-to-face survey to smokers with high-risk COPD. No other specified interventions will be given, they will be always accessible to usual care within the study period.

INTERVENTIONS:
Combination Product: Multi-component intervention for smokers — 1. Community-based spirometry pulmonary function tests and result interpretations and health education;
  2. A digital health intervention program, NicQuit, for smokers(very familiar with intelligent mobile phone);
  3. A digital health intervention program, EmoEase, for smokers whose WEMWBS questionnaire score is lower than 45(very familiar with intelligent mobile phone);
  4. Health education to smokers for smoking cessation;
  5. Health education to smokers with mental health issues;
  6. Encouragement to seek professional medication treatment in superior hospitals for spirometry-defined COPD patients or asthma patients;
  7. To actively include smokers whose blood pressure's higher than 140/90 mmHg or/and whose random blood glucose higher than11.1mmol/L into the National Essential Public Health Service in China;
  8. A CBT-based health education to the BMI abnormal, i.e., BMI > 24.0 or BMI <18.5;
  9. Pay-for-population mechanism for medical practitioners.
  Arms: Intervention arm

SUMMARY:
Study Participants: In our study, we focus on smokers who self-report a "current smoking" status or smoking cessation less than 6 months. This trial is a sub-trial of "Impact of Multi-Component Interventions on a High-Risk COPD population" (Protocol ID: CAMS&PUMC-IEC-2024-040). All smokers in this trial are either from the high-risk COPD population (defined by COPD-SQ score≥16) .

Intervention: For study participants in the intervention arm, we will ask them to finish an online COPD-SQ questionnaire with notification of his or her COPD high risk. For those whose score of COPD-SQ ≥ 16, we will provide a face-to-face survey, simple physical examination, pulmonary function tests, and provide a multi-component intervention at baseline. For smokers in the intervention arm, we provide a digital health intervention program, NicQuit, to whom could familiarly use intelligent mobile phones, and health education for all smokers. We also provide community-based spirometry pulmonary function test (PFT) and education to smokers. If smokers whose post-bronchodilator FEV1/FVC<0.7, they will be spirometry-defined COPD patients and will be encouraged to seek treatment and medication to the superior hospitals. Additionally, we provide (1) another digital health intervention programs to smokers with mental health issues; (2) CBT-based health education for study participants with abnormal BMI; (3) active recruitment into National Essential Public Health Program in China for those with abnormal blood pressure and blood glucose. Intensive follow-ups will be conducted at month 3 (telephone interview), month 6 (face-to-face with full steps of physical examination), and month 12.

Comparison: Those who are assigned in the control arm, we will ask them to finish the same COPD-SQ online questionnaire with notification of his or her COPD high risk status and a face-to-face survey. No physical examinations, community-based pulmonary function tests will be given.

Outcomes: The primary outcomes are self-reported average number of cigarettes consumed per day, smoking dependence index, and CO measurement.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 and above;
* High-risk COPD population defined by the score of COPD-SQ ≥ 16;
* Self-report currently smoking or smoking cessation less than 6 month;
* Local residents who stay within a township in the previous 3 months and plan to stay within the same township for the next 12 months.

Exclusion Criteria:

* Those who suffer from severe cognitive disorder or total loss of ability of daily living.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7400 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Amount of smoking | 1 year
  Definition: Average number of cigarettes smoked per day; Variable type: Continuous; Measurement: Respondent's answer to the question.
Smoking Dependence | 1 year
  Definition: A scale that measures the degree of smoking dependence; Variable type: Continuous; Measurement: Respondent's answer to the question. Introduction to Smoking Dependence Scale: Chinese version of Fagerström test for nicotine dependence (FTND), ranging from 0 to 15, the higher the score, the severer nicotine dependence will be. Also Heaviness of Smoking Index (HSI) will also be measured, ranging from 0 to 6, the higher the score, the worsen the nicotine dependence will be

SECONDARY OUTCOMES:
Self-rate health status | 1 year
  Definition: General self-assessed health status; Variable type: Continuous; Measurement: EQ-5D scale; Introduction to EQ-5D-5L scale: The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The scale could be transferred to health utility value, ranging from 0 to 1 continuously. 0 represents death and 1 represents perfect health.
Number of Chronic Conditions Controlled | 1 year
  Definition: Among 7 objectively measured health conditions (COPD, asthma, depression symptoms, anxiety symptoms, BMI, hypertension, type 2 diabetes), the number of chronic conditions controlled; Variable type: Counting data; Measurement: Through objective physical examination or validated scale;
Physical proof of cigarettes | 1 year
  Definition: Can you show me your cigarettes? Variable type: Binary; Measurement: Self-report questions and to let respondents show to our field workers whether he or she brings cigarettes.
FEV1 measurement | 1 year
  Definition: Forced Expiratory Volume in one second (FEV1); Variable type: Continuous; Measurement: Pulmonary function test, portable spirometry;
COPD Screening | 1 year
  Definition: Have you ever had a pulmonary function test?; Variable type: Binary; Measurement: Respondent's answer to the question;
Self-awareness of COPD | 1 year
  Definition: Have you ever been diagnosed with COPD?; Variable type: Binary; Measurement: Respondent's answer to the question;
COPD-Knowledge | 1 year
  Definition: COPD Knowledge Questionnaire; Variable type: Continuous; Measurement: Respondent's answer to the questions;
Treatment adherence | 1 year
  Definition: Are you currently receiving a COPD treatment plan prescribed by a doctor or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
COPD control | 1 year
  Definition: Has the number of acute exacerbations decreased in the past six months?; Variable type: Binary; Measurement: Respondent's answer to the question;
Blood pressure | 1 year
  Definition: Systolic and diastolic blood pressure (mmHg); Variable type: Continuous; Measurement: Omron portable automatic blood pressure monitor;
Blood Glucose | 1 year
  Definition: Reference standard for average plasma glucose concentration over a period of time; Variable type: Continuous; Measurement: Blood glucose meter;
Waist circumference | 1 year
  Definition: Waist circumference (cm); Variable type: Continuous; Measurement: Soft measuring tape;
BMI | 1 year
  Definition: Body mass index (BMI), weight divided by height squared (kg/m²); Variable type: Continuous; Measurement: Calculation;
Number of Outpatient Visits | 1 year
  Definition: Outpatient visits and type of hospital; Variable type: Count; Measurement: Survey/insurance/outpatient data;
Number of Inpatient Visits | 1 year
  Definition: Inpatient visits and type of hospital; Variable type: Count; Measurement: Survey data/insurance/inpatient data;
Medical expenditure within a family over the past year | 1 year
  Definition: Healthcare-related expenditures; Variable type: Continuous; Measurement: Survey/insurance/outpatient/inpatient data;
Depression Symptoms | 1 year
  Definition: Emotional disorders, including sadness, loss, and anger; Variable type: Continuous; Measurement: PHQ-9; Introduction to PHQ-9: Patient Health Questionnaire- 9 items (PHQ-9), ranging from 0 to 27, the higher the score, the severer the depression symptoms for the respondents will be.
Anxiety Symptoms | 1 year
  Definition: Unpleasant state of inner turmoil; Variable type: Continuous; Measurement: GAD-7; Introduction to GAD-7: General Anxiety Disorder - 7 (GAD-7), ranging from 0 to 21, the higher the score, the severer the anxiety symptoms for the respondents will be.
Warwick-Edinburgh Mental Well-being Scale, WEM -WBS | 1 year
  Definition: Reflects overall mental health problems; Variable type: Continuous; Measurement: WEMWBS; Introduction to WEMWBS: Warwick-Edinburgh Mental Well-being Scale, ranging from 14 to 70, the lower the score, the worse one's general mental health will be.
Productivity Loss | 1 year
  Definition: Productivity loss due to illness or health problems; Variable type: Continuous; Measurement: Respondent's answer to the question;
  Introduction to WPAI-GH : Work Productivity and Activity Impairment-General Health (v2.0) Chinese version.WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Questions:
  1. = currently employed
  2. = hours missed due to health problems
  3. = hours missed other reasons
  4. = hours actually worked
  5. = degree health affected productivity while working
  6. = degree health affected regular activities
  Scores:
  Multiply scores by 100 to express in percentages.
  Percent work time missed due to health: Q2/(Q2+Q4)
  Percent impairment while working due to health: Q5/10
  Percent overall work impairment due to health:
  Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)]
  Percent activity impairment due to health: Q6/10
HBP Screening | 1 year
  Definition: Have you ever had your blood pressure measured by a doctor, nurse, or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Diagnosis | 1 year
  Definition: Have you ever been diagnosed with hypertension by a doctor?; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Treatment | 1 year
  Definition: Are you currently taking any antihypertensive medication prescribed by a doctor or other healthcare professional? ; Variable type: Binary; Measurement: Respondent's answer to the question;
HBP Control | 1 year
  Definition: Blood pressure within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood pressure measurement;
T2DM Screening | 1 year
  Definition: Have you ever had your blood glucose measured by a doctor, nurse, or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Diagnosis | 1 year
  Definition: Have you ever been diagnosed with T2DM by a doctor?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Treatment | 1 year
  Definition: Are you currently receiving a type 2 diabetes treatment plan prescribed by a doctor or other healthcare professional?; Variable type: Binary; Measurement: Respondent's answer to the question;
T2DM Control | 1 year
  Definition: Blood glucose within the normal range at the end-of-year follow-up; Variable type: Binary; Measurement: Blood glucose measurement;
Smoking Status | 1 year
  Definition: Do you currently smoke?; Variable type: Binary; Measurement: Respondent's answer to the question;
Drinking Status | 1 year
  Definition: Frequency of alcohol consumption in the past 3 months; Variable type: Categorical; Measurement: Respondent's answer to the question;
Sugar Consumption | 1 year
  Definition: Frequency of consumption of sugary foods/drinks; Variable type: Categorical; Measurement: Respondent's answer to the question;
Salted Vegetables Consumption | 1 year
  Definition: Frequency of consumption of salty vegetables; Variable type: Categorical; Measurement: Respondent's answer to the question;
Vegetable Consumption | 1 year
  Definition: Frequency of consumption of vegetable; Variable type: Categorical; Measurement: Respondent's answer to the question;
Physical exercise | 1 year
  Definition: Hours of physical exercise per week; Variable type: Count; Measurement: Respondent's answer to the question;

CONTACTS AND LOCATIONS:
Overall Officials: Simiao Chen, Ph.D., Principal Investigator — Peking Union Medical College
Locations (1):
- Xishui County for Xishui Trial, Zunyi, Guizhou, China

IPD SHARING:
Plan to Share IPD: No